CLINICAL TRIAL: NCT00706004
Title: Short Term Safety and Efficacy of Lubiprostone in Adults With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Catherine E. O'Brien, University of Arkansas for Medical Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 76992
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Results first posted 2011-04-18 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-03

CONDITIONS: Constipation; Cystic Fibrosis
Keywords: constipation; cystic fibrosis; lubiprostone; Constipation in adults with cystic fibrosis
MeSH Terms: conditions — Constipation; Cystic Fibrosis | interventions — Lubiprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: lubiprostone — lubiprostone 24 microgram capsule taken twice daily for 4 weeks
  Other Names: Brand name: Amitiza

SUMMARY:
The purpose of this study is to determine the short term safety and effectiveness of lubiprostone when used for constipation in adults with cystic fibrosis.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) affects about 30,000 people in the United States. It is caused by an absent or dysfunctional protein called CF transmembrane conductance regulator (CFTR) which functions as a chloride channel. Lubiprostone is a medication indicated for constipation that activates type 2 chloride channels (ClC-2) and has the potential to be an effective treatment for constipation in adults with CF. It has the potential to correct the underlying disorder by utilizing a chloride channel whose activity does not depend on CFTR. This project is a prospective open-label pilot study to examine the safety and effectiveness of lubiprostone when used in adults with CF with constipation. The specific aims are as follows: 1) Determine the effectiveness of lubiprostone for constipation in participants with CF, and 2) Determine the short term safety of lubiprostone in adults with CF. Data will also be collected to generate further information about the effect of lubiprostone on nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of all races
* 18 years of age or older at time of enrollment
* Diagnosis of cystic fibrosis
* History of constipation, as defined by the Rome III criteria, OR the requirement of chronic scheduled doses of a laxative, OR a score ≥1.5 on the Patient assessment of constipation symptoms (PAC-SYM)15 survey administered during the screening visit, OR a score of less than 3 on the Bristol Stool Scale (BSS) at the screening visit.

Exclusion Criteria:

* Current gastrointestinal (GI) obstruction
* History of GI obstruction requiring hospitalization within six months of enrollment
* Pregnancy or breastfeeding
* Hypersensitivity to lubiprostone or any of its components
* Serum creatinine >1.8 mg/dL at last annual visit
* Clinically significant liver disease, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3X upper limit of normal
* History of frequent hospital admissions for CF exacerbations (≥4 in the last 6 months)
* Currently registered on a lung transplant waiting list
* Women of capable of child-bearing who either refuse a pregnancy test, or are incapable or unwilling to use contraception during the protocol, or both.
* Any other condition, in the opinion of the investigators, that interferes with the ability of the participant to comply with study requirements, confers significant risk to the participant, or limits the ability of the participant to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E. O'Brien, Pharm.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lubiprostone: 24 micrograms twice daily
Period: Overall Study
Arm/Group | Lubiprostone
Started | 9
Completed | 7
Not Completed | 2
Not completed — Did not meet eligibility criteria | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lubiprostone
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants] — The number of subjects analyzed here is 7 as only 7 completed this pilot study.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 7
    >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] — The number of subjects analyzed here is 7 as only 7 completed this pilot study.
  years | 26 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants] — The number of subjects analyzed here is 7 as only 7 completed this pilot study.
  Participants
    Female | 4
    Male | 3
Region of Enrollment [Number; unit: participants] — The number of subjects analyzed here is 7 as only 7 completed this pilot study.
  participants
    United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Spontaneous Bowel Movements Per Week
Time Frame: 2-week run-in period, 2-weeks of treatment, 4-weeks of treatment
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: bowel movements
Groups:
- Lubiprostone 24 Mcg Twice Daily: Participants served as their own controls
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
bowel movements
  Baseline period | 9.7 (5.7)
  2 weeks | 10.8 (5.1)
  4 weeks | 8.8 (2.9)

2. Secondary Outcome: Patient Assessment of Constipation Symptoms
Description: The Patient Assessment of Constipation - Symptom (PAC-SYM) survey is a 1-page 12-item tool that measures a patient's assessment of constipation symptoms. The items are in Likert scale format and address the severity of stool, rectal and abdominal symptoms over the past 2 weeks. Items are scored on a scale of 0 to 4, with 4 indicating the most severe. To compute the overall score, the scores of the non-missing items are summed and this is divided by the total number of non-missing items (overall score range, 0 to 4).
Time Frame: 2-week run-in period, 2 weeks of treatment, 4 weeks of treatment
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
scores on a scale
  Baseline | 1.18 (0.56)
  2 weeks | 0.54 (0.27)
  4 weeks | 0.44 (0.36)

3. Secondary Outcome: Bristol Stool Scale Score
Description: The Bristol Stool Scale is a scale used to rate the consistency of stool. Stool types are accompanied by a written description. There are seven types of stool that are scored from 1 to 7. A score of 1 or 2 indicates constipation; a score of 6 or 7, diarrhea.
Time Frame: 2-week run-in period, 2 weeks of treatment, 4 weeks of treatment
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
scores on a scale
  Baseline | 3.4 (1.1)
  2 weeks | 3.6 (0.8)
  4 weeks | 3.3 (1.1)

4. Secondary Outcome: Body Mass Index
Time Frame: baseline, 2 weeks of treatment, 4 weeks of treatment
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
kg/m^2
  Baseline | 24.0 (2.8)
  2 weeks | 24.0 (2.5)
  4 weeks | 24.3 (2.5)

5. Secondary Outcome: Self Reported Adverse Effects at Each Study Visit
Description: Adverse effects are problems reported by each study subject that they experienced during this clinical trial. Examples are headache and nausea. Study subjects were asked at each visit while on study drug to report any adverse affects that had occurred since the last visit.
Time Frame: During entire study period
Population: Participants who completed the study
Measure: Number; unit: participants
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
participants
  2 weeks | 5
  4 weeks | 3

6. Secondary Outcome: Serum Sodium
Time Frame: baseline, 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
nmol/L
  Baseline | 137.4 (2.8)
  4 weeks | 139.2 (3.6)

7. Secondary Outcome: Serum Chloride
Time Frame: baseline and 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
nmol/L
  Baseline | 103.0 (3.9)
  4 weeks | 104.3 (3.4)

8. Secondary Outcome: Serum Potassium
Time Frame: baseline and 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
nmol/L
  Baseline | 4.4 (0.4)
  4 weeks | 4.4 (0.2)

9. Secondary Outcome: Serum Bicarb
Time Frame: baseline and 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
nmol/L
  Baseline | 23.8 (4.0)
  4 weeks | 25.2 (3.3)

10. Secondary Outcome: Serum BUN
Time Frame: baseline and 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
mg/dL
  Baseline | 13.0 (4.6)
  4 weeks | 12.7 (3.3)

11. Secondary Outcome: Serum Creatinine
Time Frame: baseline and 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
mg/dL
  Baseline | 0.79 (0.15)
  4 weeks | 0.84 (0.10)

12. Secondary Outcome: AST
Time Frame: baseline and 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
U/L
  Baseline | 20.6 (11.1)
  4 weeks | 17.5 (3.9)

13. Secondary Outcome: ALT
Time Frame: baseline and 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
U/L
  Baseline | 25.1 (16.7)
  4 weeks | 23.8 (14.5)

14. Secondary Outcome: Serum Calcium
Time Frame: baseline and 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
mg/dL
  Baseline | 9.3 (0.3)
  4 weeks | 9.3 (0.2)

15. Secondary Outcome: Serum Magnesium
Time Frame: baseline and 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
mg/dL
  Baseline | 2.0 (0.3)
  4 weeks | 2.0 (0.2)

16. Secondary Outcome: Serum Phosphate
Time Frame: baseline and 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
mg/dL
  Baseline | 3.8 (0.6)
  4 weeks | 3.7 (0.5)

17. Secondary Outcome: Serum Glucose
Time Frame: baseline and 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
mg/dL
  Baseline | 150.3 (101.9)
  4 weeks | 131.8 (83.3)

18. Secondary Outcome: Serum Vitamin D
Time Frame: baseline and 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
ng/mL
  Baseline | 25.3 (15.9)
  4 weeks | 25.3 (18.4)

19. Secondary Outcome: Serum Vitamin A
Time Frame: baseline and 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
ug/dL
  Baseline | 41.3 (14.6)
  4 weeks | 42.7 (23.3)

20. Secondary Outcome: Serum Vitamin E
Time Frame: baseline and 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
mg/L
  Baseline | 6.6 (3.4)
  4 weeks | 7.7 (6.1)

21. Secondary Outcome: Serum Prealbumin
Time Frame: baseline and 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
mg/dL
  Baseline | 22.6 (3.3)
  4 weeks | 21.5 (6.1)

22. Secondary Outcome: Serum Albumin
Time Frame: baseline and 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Lubiprostone 24 Mcg Twice Daily
Number analyzed (Participants) | 7
g/dL
  Baseline | 4.3 (0.3)
  4 weeks | 4.3 (0.2)

ADVERSE EVENTS:
Arm/Group | Lubiprostone
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 6/7
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lubiprostone (N=7)
Nausea (Gastrointestinal disorders) | 2 (3)
Abdominal bloating (Gastrointestinal disorders) | 1 (1)
Abdominal cramping (Gastrointestinal disorders) | 1 (2)
Heartburn (Gastrointestinal disorders) | 1 (1)
Headache (General disorders) | 1 (2)
Migraine (General disorders) | 1 (1)
Insomnia (General disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Transient chest tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes